CLINICAL TRIAL: NCT05367245
Title: Microbiome Targeted Oral Butyrate Therapy in Gulf War Multisymptom Illness
Brief Title: Ca-Mg Butyrate in GWI
Acronym: Butyrate
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Miami VA Healthcare System (U.S. Federal Agency); VA Salt Lake City Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPLD-006-21S; I01CX002372 (NIH)
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Gulf War Illness; Chronic Fatigue; Neurocognitive Dysfunction
Keywords: SCFA; Gulf War Illness; GWI; Microbiome; Butyric acid; Butyrate
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Intervention Model Description: -Drug: Ca-Mg-Butyrate Take oral Capsule as directed (600 mg, two times a day for 18 weeks; 2x600 mg/day for 18 weeks) with food or without food.
  Other name: Calcium-Magnesium Butyrate, BodyBio Cal-Mag Butyrate
  -Drug: Placebo Take oral Capsule as directed (600 mg, two times a day for 18 weeks; 2x600 mg/day for 18 weeks) with food or without food.
  Other Name: Sugar pill, inactive substance
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple, participants, care provider, investigators and outcome assessor will not have access to blinding. Only research pharmacist to distribute the drug or placebo and study coordinator to keep a confidential and secure records, will have access to the blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cal-Mag-Butyrate (Experimental): Take oral capsule as directed (600 mg, twice a day for 18 weeks) with or without food.
  Interventions: Drug: Cal-Mag Butyrate
- Placebo for Cal-Mag-Butyrate (Placebo Comparator): Take oral capsule as directed (600 mg, twice a day for 18 weeks) with or without food.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cal-Mag Butyrate — Supplements
  Other Names: Bodybio Calcium Magnesium Butyrate
  Arms: Cal-Mag-Butyrate
Drug: Placebo — Only Cal-Mag but no Butyric acid
  Other Names: Placebo Cal-Mag Butyrate
  Arms: Placebo for Cal-Mag-Butyrate

SUMMARY:
The primary objective of this clinical trial is to determine if treatment with Butyrate formulation that consists of butyric acid as calcium and magnesium derivatives (Ca-Mg Butyrate) improves the physical function of men and women Veterans suffering from Gulf War Illness (GWI). The primary outcome measure is a change from baseline on the Short Form Health Survey 36-item (VSF-36), with respect to physical functioning and symptoms. The secondary outcome will focus on the drug's role in (a) restoring gut microbiome and virome, (b) decreasing gastrointestinal disturbances (constipation, diarrhea, pain), (c) decreasing chronic fatigue, (d) decreasing systemic inflammation, and (e) a decrease in cognitive deficits.

DETAILED DESCRIPTION:
Nearly one third of 700,000 military personnel deployed during Desert Shield and Desert Storm (Aug 2, 1990 to July 31, 1991) in the Kuwaiti War Theater are suffering from Gulf War Illness (GWI), an unexplained chronic illness characterized by multiple symptoms. The illness has taken a heavy toll on deployed Veterans' overall quality of life. Recent research has revealed the host gut microbiome's role in gastrointestinal disturbance, systemic inflammation, and neurotrophic abnormalities in Gulf War Illness mouse models. Also, short-chain fatty acids such as butyrate restored a healthy microbiome and improved gut microbial metabolism apart from attenuating GWI symptom persistence in preclinical studies. Butyrate, a nutraceutical endogenously produced in the host gut following bacterial fermentation, has shown promise in gastrointestinal disturbances such as irritable bowel syndrome (IBS) and Inflammatory bowel disease (IBD).

This is a randomized, two-group, double-blind, placebo-controlled, Phase II clinical trial. The treatment group will receive microencapsulated butyrate capsules (600 mg twice a day for 18 weeks). The placebo group will receive a matching placebo formulation twice a day for 18 weeks. However, after two weeks of the treatment (20 weeks) there will be a follow up virtual visits. The primary outcome measure for this clinical trial is a change from baseline of VSF-36 and CVLT III test scores with respect to physical and mental functioning and symptoms. The secondary outcome measures include changes from baseline of host-microbiome signature, intestinal permeability assessment, peripheral pro-inflammatory biomarkers, and GWI-associated symptoms IBS, chronic pain, fatigue, sleep issues, and cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Gulf war era veteran deployed 40 and 70 years old, in good health by medical history prior to 1990 meeting GWI case definition of CDC and Kansas criteria and
* currently have no exclusionary diagnoses (self- reported) that could reasonably explain the symptoms of their fatiguing illness. The severity of illness is moderate to severe, scoring less than 30 of 100 on the physical domain of VSF36 .

Exclusion Criteria:

* Untreated schizophrenia,
* Untreated bipolar disorder,
* Untreated delusional disorders,
* Untreated dementias of any type and
* active alcoholism or drug abuse.
* Medical conditions excluded include (i) organ failure, (ii) defined rheumatologic inflammatory disorders, and (iii) transplant.
* Use of Butyrate in any form in the 3 months prior to study drug, medications that would impact gut motility, diarrhea, chronic pain, and immune function e.g., steroids, (Last 3 months)
* immunosuppressive drugs or biologic response modifiers within 3 months of study entry will be used as exclusion criteria.
* Pregnancy, or planned pregnancy in the next 6 months,
* Body mass index more than 35
* Specific diets that may have enhanced or enriched fiber or butyrogenic formulations (FODMAP)
* Medications that could potentially impact immune function in the past one month will be excluded (e.g., steroids, antibiotics, immunosuppressives;
* Medications containing supplement calcium or magnesium butyrate should not be taken for at least 3 months before study entry.
* Nutraceuticals that are formulated to impact gut microbiome or immune health) and use of drugs that affect GI motility and use of any antibiotic in the last 2 months.
* Known allergy to butyrate supplements or their derivatives such as sodium salts or hydroxy derivatives of butyrate and/or inactive ingredients of active and placebo soft gelatin will also be excluded.
* Current evidence of celiac disease or late-stage cirrhosis of the liver, Giardia antigen presence, Clostridium difficile toxin in stool, tissue transglutaminase antibody, recent change in gastrointestinal medications, use of drugs that affects gastrointestinal motility, and use of any antibiotic in the last two months also will be excluded.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-10-10 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Veterans Short Form 36-Item Health Survey Physical Component Summary | Change from Baseline at 3, 6, 9, 12, 18 and 20 weeks
  Veterans Health Survey contains 36 items to measure health functioning from the patient's point of view. Qualify of life will be determined per Short Form-36 for Veterans' quality of life Physical component (PCS) summary scales, range from 0 to 100 with 100 being better; 50 is expected population average.

SECONDARY OUTCOMES:
California Verbal Learning Test (CVLT-II) | Change from Baseline at 9, 18 and 20 weeks
  CVLT-II asks questions about cognitive symptoms related to recall and memory. The CVLT-II is used to measure verbal learning and episodic long-term memory. It assesses learning, short- and long-delayed recall and recognition for a list of 16 shopping items. Subjects are expected to remember a list of words. They are asked to repeat the words remembered 5 times (5 trials). Each of the words correctly remembered, in each trial, is marked as 1 point. The reported data represent the number of correct items for the Trial 1-Trial 5, Short Delay Free Recall, and Long Delay Free Recall. The long-delayed recall is assessed at 20 minutes. The CVLT enables a comprehensive characterization of a participant's memory profile. Scale ranges from 0 to 80 with 80 being the best.

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh Chatterjee, PhD, Principal Investigator — VA Long Beach Healthcare System, Long Beach, CA
Locations (3):
- United States (3):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No